CLINICAL TRIAL: NCT00782366
Title: Proof-of-Principle Trial of Communication to Patients Receiving Predictive Genetic Risk Assessment
Brief Title: Predictive Genetic Risk Assessment Trial
Acronym: PGT
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Clayton T. Cowl, M.D., Mayo Clinic
Other Study IDs: 07-007414
Record Dates: First submitted 2008-10-29; First posted 2008-10-31 (Estimated); Last update posted 2011-04-27 (Estimated); Status verified 2011-04

CONDITIONS: Colon Cancer; Lung Cancer; Atrial Fibrillation; Diabetes Type 2; Obesity; Breast Cancer; Graves Disease; Osteoarthritis; Celiac Disease; Myocardial Infarction; Prostate Cancer
Keywords: predictive genomics; personalized medicine; personal genomics; direct-to-consumer genetic testing; genetic knowledge; genetic attitudes
MeSH Terms: conditions — Colonic Neoplasms; Lung Neoplasms; Atrial Fibrillation; Diabetes Mellitus, Type 2; Obesity; Breast Neoplasms; Graves Disease; Osteoarthritis; Celiac Disease; Myocardial Infarction; Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Genetic Testing Group: Those who will receive predictive genetic risk assessments
  Interventions: Genetic: SNP analysis
- Control: Those who will receive standard of care

INTERVENTIONS:
Genetic: SNP analysis — The patients in the intervention group will obtain genetic risk assessments based on genome-wide association studies.
  Other Names: Navigenics
  Groups: Genetic Testing Group

SUMMARY:
This proof-of-principle clinical trial at Mayo Clinic studies how patients and their physicians understand and utilize predictive genetic risk assessment. A critical goal of this clinical trial is to understand how individual patients and their doctors perceive and respond to genetic risk information that is largely uncertain.

DETAILED DESCRIPTION:
The prospect of personalized medicine is under heated debate at the Mayo Clinic and it is of interest across the world. A point of contention is the provision of individual genetic risk assessment to healthy patients, especially information predicting risk of common diseases like diabetes, cancer, or heart disease. While scientific debate continues, personal genetic testing is currently offered to the public by commercial firms using a "direct-to-consumer" (DTC) approach. At present, the number of private companies offering such services is growing (i.e. 23 and me, deCode genetics, etc.). Although many professionals hope that genetic risk information will prove to be valuable in the near future, there is little understanding of how this kind of predictive risk assessment will be interpreted and perceived by patients and their doctors. Due to the great attention given to predictive genetic testing in the popular press, one expects that patients will soon demand this testing as part of standard clinical practice. Yet, there is currently no effective regulatory oversight to guide clinicians and policy makers about how to incorporate results from predictive genetic testing into routine clinical use. In fact, no appropriate clinical trials assessing the impact of this type of testing have been completed. Indeed, a recent commentary in the New England Journal of Medicine recommended that all such testing be conducted in the context of a clinical trial.

How to protect human subjects during the early stages of development of a new technology is a classic dilemma in translational research. For that reason, we have developed a "proof-of-principle" clinical trial at Mayo Clinic to study how patients and their physicians understand and utilize predictive genetic risk assessment. A critical goal of this clinical trial is to understand how individual patients and their doctors perceive and respond to genetic risk information that is largely uncertain.

Our pilot study seeks to answer three fundamental questions: How will physicians deal with the uncertainty provided by the new technology of predictive genetic risk assessment? What hopes do patients have regarding the significance of predictive genetic testing? And how do they interpret their results? This proof-of-principle study will investigate the impact of direct-to-consumer, predictive genetic testing provided and sponsored by Navigenics, Inc., a private company advertising predictive genetic testing for common diseases or conditions. This study will allow Mayo Clinic to be proactive in researching the dynamics of this potential innovation in health care. The proof-of-principle study described herein is designed to collect preliminary data that will inform the development of a larger clinical trial and provide data for an application for federal funding.

Our study will be in collaboration with Navigenics, the industry sponsor of this project. Navigenics will use a high density, genome microarray for determining the gene variants-, and published disease-association studies, to calculate the relative risk of each patient for a few targeted common diseases. High density microarrays are genome chips that allow the assessment of one million single nucleotide polymorphisms (SNPs) at relatively low cost. The combination of particular SNPs are presumed to influence the risk of developing certain common diseases as shown from genome-wide association studies published in peer-reviewed scientific and medical literature. Navigenics will use these population-based association studies (studies that produce odds ratios for developing a disease given a certain SNP) to estimate the relative of an individual patient developing a disease, an approach that is used by most direct-to-consumer genetic testing companies. They claim that their testing has a role in preventive medicine in order to "Help people live healthier lives." Our study will allow us to examine how patients and doctors respond to and utilize Navigenics' risk assessments derived from microarray technology and published genome-wide association studies.

The role of information delivery to patients by physicians, genetic counselors or other health care professionals using predictive genetic risk assessment is unclear. Its acceptance by patients and health care professionals has also not been studied. Therefore, this study seeks to compare the perception of genetic risk estimations obtained from Navigenics' testing with the relative risk estimations obtained through a family history, the current Mayo standard of care.

Our study design includes two phases to be conducted over 18 months. The first phase is a "pre-pilot" study that will take place in 2008. In phase one, we will conduct structured interviews with 20 Executive Health (EH) Program patients who have obtained their disease risk assessments for common diseases or who have obtained a family history. In phase 2, we will conduct a quantitative phone survey with 150 EH patients randomized into two arms (genetic testing and standard of care). We will also conduct follow up qualitative interviews with 20 patients in phase 2. The study is anticipated to be completed in mid 2009.

ELIGIBILITY:
Inclusion Criteria:

* must be established EH patient or physician

Exclusion Criteria:

* pregnant women
* patient who have already purchased Navigenics Health Compass

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients and physicians from the Mayo Clinic Rochester Executive Health (EH) program will be recruited to participate in this study
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2008-03; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Assess accessibility and feasibility, including positive and negative aspects of integrating predictive genomics at the clinic focusing on patients' and physicians' attitudes | March 2008-March 2009

SECONDARY OUTCOMES:
Assess effects of predictive genomics on self-reported health behavior and on physician-patient interaction | March 2008-March 2009

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Tiedje, Ph.D., Study Director — Mayo Clinic; Clayton T. Cowl, M.D., Principal Investigator — Mayo Clinic; Barbara A. Koenig, Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] James KM, Cowl CT, Tilburt JC, Sinicrope PS, Robinson ME, Frimannsdottir KR, Tiedje K, Koenig BA. Impact of direct-to-consumer predictive genomic testing on risk perception and worry among patients receiving routine care in a preventive health clinic. Mayo Clin Proc. 2011 Oct;86(10):933-40. doi: 10.4065/mcp.2011.0190. PMID 21964170